CLINICAL TRIAL: NCT06167967
Title: Circulating Tumor DNA Methylation Guiding Postoperative Adjuvant Chemotherapy in Stage III Colorectal Cancer: a Multicenter, Randomized Controlled Trial
Brief Title: Circulating Tumor DNA Methylation Guiding Postoperative Adjuvant Chemotherapy in Stage III Colorectal Cancer
Acronym: cmPAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Zhangfa Song, Vice director, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SRRS-cmPAT; SRRS2023-0704 (Registry Identifier: Ethics Committee of Sir Run Run Shaw Hospital, School of Medicine)
Record Dates: First submitted 2023-12-04; First posted 2023-12-13 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; ctDNA methylation; adjuvant chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ctDNA-guided group (Experimental): ctDNA-negative group in the high-risk cohort were treated with XELOX regimen for 6 months; ctDNA-positive group in the high-risk cohort was treated with cmFOLFOXIRI regimen for 6 months; ctDNA-positive group in the low-risk cohort were treated with XELOX regimen for 3 months; ctDNA-negative group in the low-risk cohort did not receive adjuvant chemotherapy.
  Interventions: Diagnostic Test: ctDNA methylation
- standard treatment group (Active Comparator): The standard treatment group in the high-risk cohort were treated with XELOX regimen for 6 months, and in the low-risk cohort were treated with XELOX regimen for 3 months.
  Interventions: Diagnostic Test: standard treatment

INTERVENTIONS:
Diagnostic Test: ctDNA methylation — A blood-based circulating tumor DNA methylation assay that uses 6 different methylation markers, SEPT9 region1, SEPT9 region2, BCAT1, IKZF1, BCAN and VAV3.
  Arms: ctDNA-guided group
Diagnostic Test: standard treatment — This group was treated according to standard procedure
  Arms: standard treatment group

SUMMARY:
The goal of this randomized controlled trial is to investigate whether ctDNA methylation is a more precise indicator to guide postoperative adjuvant chemotherapy in stage Ill colorectal cancer. The main questions it aims to answer are:

1. Whether ctDNA methylation-guided escalation strategy is superior to standard treatment for stage III high-risk CRC patients.
2. Whether ctDNA methylation-guided de-escalation strategy is non-inferior to standard treatment for stage III low-risk CRC patients.

325 cases were included in the high-risk cohort (T4 and/or N2) and 665 cases were included in the low-risk cohort (T1-T3, N1). Then patients in each cohort were randomly assigned to ctDNA-guided treatment (ctDNA-guided group) and standard treatment (standard treatment group) in a ratio of 2:1. The standard treatment group and ctDNA-negative group in the high-risk cohort were treated with XELOX regimen for 6 months, and the ctDNA-positive group in the high-risk cohort was treated with cmFOLFOXIRI regimen for 6 months. The standard treatment group and the ctDNA-positive group in the low-risk cohort were treated with XELOX regimen for 3 months, while the ctDNA-negative group in the low-risk cohort did not receive adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old ≤ age < 75 years old.
2. Stage III (T1-4, N1-2, M0) colorectal cancer patients.
3. Patients who can undergo R0 resection.
4. ECOG score 0 ~ 2.
5. Expected survival ≥ 6 months.
6. No history of other malignant tumors.
7. Voluntarily participate in this study and sign the informed consent. If the subject does not have the ability to read the informed consent (e.g., illiterate subjects), a witness must witness the informed process and sign the informed consent.

Exclusion Criteria:

1. Patients who have received neoadjuvant chemotherapy.
2. Known high clinical risk of adjuvant chemotherapy.
3. Patients with clear contraindications to adjuvant chemotherapy (i.e. due to physical condition, comorbidities, active second cancer, or age).
4. Patients who are unable to undergo subsequent chemotherapy due to other reasons (travel distance, compliance).
5. Vulnerable groups, including people with mental illness, people with cognitive impairment, critically ill patients, minors, pregnant women, etc.
6. There are any other circumstances that the researcher deems unsuitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 990 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival at 3 years | 3 years

SECONDARY OUTCOMES:
Overall survival at 5 years | 5 years
ctDNA clearance rate in ctDNA-positive patients treated with adjuvant chemotherapy | 6 months
The proportion of patients in the low-risk cohort who did not receive adjuvant chemotherapy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhangfa Song, Dr, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shao hospital, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided